CLINICAL TRIAL: NCT03123133
Title: Gene Expression That Predicts Radiation Exposure in Humans
Status: Completed | Type: Observational
Sponsor: DxTerity Diagnostics (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: DXT-RBT-AB01
Record Dates: First submitted 2017-04-13; First posted 2017-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Total Body Irradiation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood for genomic analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To verify and validate a biodosimetry test for determining absorbed ionizing radiation dose by analyzing gene expression signatures of blood samples collected from patients treated with Total Body Irradiation (TBI).

DETAILED DESCRIPTION:
In order validate the performance of DxTerity's Radiation Biodosimetry Test (RBT) system, several clinical centers will provide controlled, de-identified blood samples and associated clinical information to DxTerity Diagnostics (DxTerity). Variations in dose and frequency of delivery in TBI protocols are expected between the clinical centers and this has been accounted for in the study design. Samples from up to 200 participants will be collected via this protocol. Blood samples for this study will be collected from radiation therapy patients receiving TBI as part of a therapeutic regimen from the site.

Blood samples (up to 4 mL per time point) may be obtained at the time of routine blood collection; participation in this biomarker study will not affect any aspect of patient treatment. Study samples will be obtained prior to, during, and post-radiation treatment regimen. Associated clinical information will be collected from the subject's medical record, as well.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients age 2 or older.
2. Weigh at least 13kg (30lbs), and in the opinion of the investigator, are healthy enough to participate in study activities.
3. Evidence of a personally signed and dated informed consent/assent document indicating that the subject or a legally acceptable representative (parent(s)/legal guardian) has been informed of all pertinent aspects of the study.
4. Diseases treated with HSCT, including malignant and nonmalignant diseases.
5. Planned fractionated total body irradiation (TBI) as part of clinical care with a cumulative dose ≥6 Gy or a single dose between 1.5 and 3.0 Gy.

Exclusion Criteria:

1. Subjects who have received chemotherapy within 21 days prior to TBI.
2. Concurrent chemotherapy with Fludarabine or an investigational product
3. Cytokine inhibitor or cytokine-inducer therapy within 30 days prior to and during the irradiation regimen
4. Subjects who have received GCSF within 30 days prior to TBI
5. Participants, who in the opinion of the investigator, may not be able to comply with the requirements of the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Blood samples for this study will be collected from radiation therapy patients receiving TBI as part of a therapeutic regimen from the site. Fractionated TBI treatment will provide a cumulative dose ≥6.0 Gy depending on the specific treatment protocol, or a single non-fractionated dose between 1.5 and 3.0 Gy.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
Collection of a sufficient number of blood samples to enable clinical validation of the RBT | Up to approximately 1 month, from informed consent through completion of blood sample and data collection activities
  Obtain blood samples from 200 TBI patients to analytically validate the Radiation Biodosimetry Test (RBT) System using peripheral blood samples. The RBT should be able to estimate the amount of absorbed radiation that an individual has received from 0 to 10 Gy for up to 7 days post-exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Aviva Jacobs, PhD, Study Director — Director, Product Developement
Locations (3):
- United States (3):
  - City of Hope, Duarte, California
  - University of California, Los Angeles, Radiation Oncology, Los Angeles, California
  - Fred Hutch Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No